CLINICAL TRIAL: NCT03635827
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Xenon Inhalation for Treatment of Patients With Posttraumatic Stress Disorder
Brief Title: Xenon Inhalation for Treatment of Posttraumatic Stress Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nobilis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBTX-001
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBTX-001 (Active Comparator)
  Interventions: Combination Product: NBTX-001 Xenon Inhaler
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: NBTX-001 Xenon Inhaler — The NBTX-001 medical gas consists of 30% xenon, 30% oxygen, and 40% nitrogen. The dose of medical gas is 10 L by volume.
  Arms: NBTX-001
Combination Product: Placebo — The placebo medical gas consists of 30% oxygen and 70% nitrogen.The dose of placebo medical gas is 10 L by volume.
  Arms: Placebo

SUMMARY:
This study is a double-blind, randomized, placebo-controlled, clinical trial in parallel groups in patients with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a current diagnosis of PTSD (documented diagnosis of PTSD based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition [DSM-5] criteria and a Clinician Administered PTSD Scale [CAPS-5] total severity score of >30).
* Male and female patients between the ages of 18 and 85 years.

Exclusion Criteria:

* History of schizophrenia, bipolar and other psychotic disorders.
* Patients with underlying pulmonary disease, chronic obstructive pulmonary disease (COPD), asthma or any other respiratory conditions / diseases that may affect the respiratory function.
* Currently undergoing PTSD-targeted psychotherapy.
* Currently undergoing exposure-based psychotherapy for any condition.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
CAPS-5 | Baseline to Week 6
  Change in CAPS-5 score

SECONDARY OUTCOMES:
PCL-5 | Baseline to Week 6
  Change in PCL-5 score

IPD SHARING:
Plan to Share IPD: Undecided